CLINICAL TRIAL: NCT05051462
Title: Efficacy of Family / Systemic Constellation Therapy in the General Population. A Randomized Wait-list Controlled Trial
Brief Title: Efficacy of Family Constellations in the General Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Károli Gáspár University of the Reformed Church in Hungary (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTK/591-1/2021
Record Dates: First submitted 2021-07-09; First posted 2021-09-21 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Mild to Moderate Psychopathological Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Study participants participating in family constellation therapy between assessment 1 and 2.
  Interventions: Behavioral: Family / systemic constellation therapy
- Wait-list control group (No Intervention): Study participants participating in family constellation therapy only after all 3 assessment points.

INTERVENTIONS:
Behavioral: Family / systemic constellation therapy — Family / systemic constellation therapy is a short-term group counseling intervention aiming to help clients better understand and resolve their conflicts within their personal systems, which in turn might lead to a decrease in psychopathological or functional somatic symptoms. The personal system addressed is most often the family but other inter- or intrapersonal systems (e.g., ego parts, victim-perpetrator dyads) can also be the target of the intervention.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate the efficacy of systemic / family constellation therapy in improving mild-moderate psychopathological symptoms and overall wellbeing in the general population. Given the limited amount of evidence on this therapeutic method, special attention will be given to monitor potential adverse outcomes to establish intervention safety. The study will use a randomized, wait-list controlled design and a 6-month follow-up time. This is the second study of this nature following a similar study from Germany.

DETAILED DESCRIPTION:
Family/systemic constellation therapy is a system-oriented, short-term group counseling intervention aiming to help clients better understand and resolve their conflicts within their intra- or interpersonal systems, which in turn might lead to a decrease in psychopathological and functional somatic symptoms as well as improvement in overall quality of life. This intervention modality was developed in Germany in the early 1990s integrating elements of - among others - psychodrama, family sculptures, contextual therapy, and certain South-African aboriginal traditions.

Compared to its widespread use by therapists of various theoretical and professional backgrounds all over the world, little effort has been made to generate empirical data regarding the efficacy and safety of this intervention and the overall quality and quantity of the extant evidence is low. Authors of the only (although high-quality) previous randomized controlled trial to date into the efficacy of systemic constellations reported that the intervention was efficacious in reducing general, non-diagnosis-specific psychopathology and psychological distress both in the short- as well as middle- and long term. A recent systematic review summarizing both the peer-reviewed and the grey literature on the mental health effects of systemic constellation therapy concluded that further studies into its efficacy and effectiveness are greatly needed, especially if employing 1) a controlled, ideally randomized-controlled design, 2) at least mid-term follow-up (≥6 months) to evaluate client outcomes and 3) active monitoring of potential iatrogenic effects.

In line with these recommendations, the aim of the present study - when designed - was to collect and analyze further data on the efficacy of systemic constellation therapy in its traditional format in improving mental health. However, the COVID pandemic required the intervention providers to make substantial changes to the usual treatment protocol; therefore, the study in its final form rather serves the purpose of investigating the efficacy of a pandemic-adjusted version of family/systemic constellation workshops than that of the intervention in general.

ELIGIBILITY:
Inclusion Criteria:

* Ability to participate in the in-person intervention on the date randomly assigned to them

Exclusion Criteria:

* Participation in family / systemic constellation therapy within the 12 months prior to study launch
* Current mental disorder diagnosed by an eligible health care professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barna Konkoly-Thege, PhD, Principal Investigator — University of Toronto
Locations (1):
- Károli Gáspár University of the Reformed Church in Hungary, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
The authors are concerned that making individual participant data available to others would seriously jeopardize participants' willingness to participate in the study.
  Therefore, the authors offer that they will conduct any alternative analyses on the data set other researchers are interested in and the authors will share the raw output of those analyses including the analytical syntaxes.

REFERENCES:
- [Background] Konkoly Thege B, Petroll C, Rivas C, Scholtens S. The Effectiveness of Family Constellation Therapy in Improving Mental Health: A Systematic Review. Fam Process. 2021 Jun;60(2):409-423. doi: 10.1111/famp.12636. Epub 2021 Feb 2. PMID 33528854
- [Background] Weinhold J, Hunger C, Bornhauser A, Link L, Rochon J, Wild B, Schweitzer J. Family constellation seminars improve psychological functioning in a general population sample: results of a randomized controlled trial. J Couns Psychol. 2013 Oct;60(4):601-9. doi: 10.1037/a0033539. Epub 2013 Aug 19. PMID 23957767
- [Result] Konkoly Thege B, Szabo GS. The efficacy of pandemic-adjusted family/systemic constellation therapy in improving psychopathological symptoms: A randomized controlled trial. J Psychiatr Res. 2024 Sep;177:271-278. doi: 10.1016/j.jpsychires.2024.07.027. Epub 2024 Jul 18. PMID 39053295

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Wait-list Control Group
Started | 37 (Out of the 37 participants of the intervention group, one participant withdrew their consent between study enrollment and baseline data collection. Therefore, we only had baseline data for 36 individuals from the intervention group.) | 43 (40 individuals were allocated to both treatment arms. However, 3 participants randomized to the intervention group were sick during the time of intervention and so did not receive the intervention and became part of the waitlist control group (in the per protocol analyses))
Completed | 35 | 33 (2 individuals were excluded due to severe protocol violation (participated in target intervention outside of the study context during the study period))
Not Completed | 2 | 10
Not completed — Lost to Follow-up | 1 | 8
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Wait-list Control Group | Total
Number analyzed (Participants) | 36 | 43 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (8.2) | 42.0 (9.9) | 42.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hungary | 36 | 43 | 79
General Severity Index of the Brief Symptom Inventory [Mean (Standard Deviation); unit: scores on a scale] — The Brief Symptom Inventory is a a broad-spectrum measure of psychopathology covering 9 symptom dimensions: Somatization, Obsessive-compulsive symptoms, Interpersonal sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation, and Psychoticism. The BSI includes a global index of distress (the General Severity Index, GSI) that reflects the mean of all items, which is used here. The GSI ranges between 0 to 4, higher scores indicative of a higher degree of symptom severity.
  scores on a scale | 0.79 (0.49) | 0.87 (0.68) | 0.83 (0.60)
Eating disorder risk assessed by the SCOFF Screening Test [Mean (Standard Deviation); unit: scores on a scale] — The SCOFF consists of five yes-or-no type questions assessing eating disorder symptoms or risk factors. Higher scores (ranging between 0 and 5) are indicative of greater risk. At least two positive answers (score of 2) indicate a high likelihood of an eating disorder.
  scores on a scale | 0.64 (0.93) | 0.75 (1.13) | 0.72 (1.05)
Substance- and behavioral addiction severity assessed by the SSBA-G [Mean (Standard Deviation); unit: scores on a scale] — The SSBA-G (Generalised version of the Screener for Substance and Behavioural Addictions) is comprised of 8 items (4 items assessing substance-related and 4 assessing behavioral addictions). Items reflect a distinct sign or symptom of potentially problematic involvement into an addictive behavior ("I did it too much;" "Once I started, I couldn't stop;" "I felt I had to do it in order to function;" and "I continued to do it, even though it caused problems"). Scores range between 8 and 56 with higher scores indicative of higher problem severity.
  scores on a scale | 12.97 (5.76) | 16.98 (11.43) | 15.33 (9.73)
Quality of life specific to interpersonal relationships assessed by the EXIS.pers [Mean (Standard Deviation); unit: scores on a scale] — The EXIS.pers assesses the subjective experiences of the individual in their personal social system (e.g. family, circle of friends) covering four dimensions in relation to belonging, autonomy, accord, and confidence. Scores range between 12 and 72 with higher scores are indicative of better functioning.
  scores on a scale | 4.06 (0.77) | 4.24 (0.87) | 4.12 (0.82)
Perceived level of meaning in life assessed by the Meaning in Life Questionnaire (MLQ) [Mean (Standard Deviation); unit: scores on a scale] — The Presence of Meaning Subscale of the MLQ assesses perceived level of meaningfulness in a respondent's life. The subscale consists of 5 items, and the total scores range between 5 and 35. Higher scores are indicative of better functioning and quality of life.
  scores on a scale | 21.03 (7.93) | 24.73 (8.60) | 23.16 (8.35)
Life satisfaction assessed by the Satisfaction With Life Scale (SWLS) [Mean (Standard Deviation); unit: scores on a scale] — The SWLS is a measure of general satisfaction with one's life. Scores range from 5 to 35 with higher scores indicative of higher life satisfaction.
  scores on a scale | 20.33 (5.17) | 21.33 (7.49) | 21.01 (6.41)
General well-being assessed by the 5-item Version of the WHO Wellbeing Index (WBI-5) [Mean (Standard Deviation); unit: scores on a scale] — The WBI-5 measures participants' overall subjective well-being. Scores range between 0 and 15 with higher scores indicative of greater well-being.
  scores on a scale | 8.33 (3.13) | 8.98 (3.24) | 8.59 (3.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Symptom Inventory Scores
Description: The Brief Symptom Inventory is a a broad-spectrum measure of psychopathology covering 9 symptom dimensions: Somatization, Obsessive-compulsive symptoms, Interpersonal sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation, and Psychoticism. The BSI includes a global index of distress (the General Severity Index, GSI) that reflects the mean of all items, which is used here. The GSI ranges between 0 to 4, higher scores indicative of a higher degree of symptom severity.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 0.61 (0.36) | 0.71 (0.68)

2. Primary Outcome: Change in Brief Symptom Inventory Scores
Description: The Brief Symptom Inventory is a a broad-spectrum measure of psychopathology covering 9 symptom dimensions: Somatization, Obsessive-compulsive symptoms, Interpersonal sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation, and Psychoticism. The BSI also includes a global index of distress (the General Severity Index, GSI) that reflects the mean of all items, which is used here. The GSI ranges between 0 to 4, higher scores indicative of a higher degree of symptom severity.
Time Frame: 6 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 33
score on a scale | 0.65 (0.40) | 0.77 (0.70)

3. Secondary Outcome: Change in Eating Disorder Risk Assessed by the SCOFF Screening Test
Description: The SCOFF consists of five yes-or-no type questions assessing eating disorder symptoms or risk factors. Higher scores (ranging between 0 and 5) are indicative of greater risk. At least two positive answers (score of 2) indicate a high likelihood of an eating disorder.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 0.66 (0.87) | 0.56 (0.89)

4. Secondary Outcome: Change in Eating Disorder Risk Assessed by the SCOFF Screening Test
Description: as for outcome 3
Time Frame: 6 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 0.66 (0.76) | 0.55 (0.90)

5. Secondary Outcome: Change in Substance- and Behavioral Addiction Severity Assessed by the SSBA-G
Description: The SSBA-G (Generalised version of the Screener for Substance and Behavioural Addictions) is comprised of 8 items (4 items assessing substance-related and 4 assessing behavioral addictions). Items reflect a distinct sign or symptom of potentially problematic involvement into an addictive behavior ("I did it too much;" "Once I started, I couldn't stop;" "I felt I had to do it in order to function;" and "I continued to do it, even though it caused problems"). Scores range between 8 and 56 with higher scores indicative of higher problem severity.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 13.83 (6.48) | 14.06 (7.92)

6. Secondary Outcome: Change in Substance- and Behavioral Addiction Severity Assessed by the SSBA-G
Description: as for outcome 5
Time Frame: 6 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 33
score on a scale | 12.71 (7.83) | 16.39 (10.97)

7. Secondary Outcome: Change in Quality of Life Specific to Interpersonal Relationships Using the Experience in Personal Social Systems Questionnaire (EXIS.Pers)
Description: The EXIS.pers assesses the subjective experiences of the individual in their personal social system (e.g. family, circle of friends) covering four dimensions in relation to belonging, autonomy, accord, and confidence. Scores range between 12 and 72 with higher scores are indicative of better functioning.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 4.13 (0.72) | 4.29 (0.84)

8. Secondary Outcome: Change in Quality of Life Specific to Interpersonal Relationships Using the Experience in Personal Social Systems Questionnaire (EXIS.Pers)
Description: as for outcome 7
Time Frame: 6 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 33
score on a scale | 4.20 (0.84) | 4.33 (0.99)

9. Secondary Outcome: Change in Perceived Level of Meaning in Life Using the Meaning in Life Questionnaire (MLQ)
Description: The Presence of Meaning Subscale of the MLQ assesses perceived level of meaningfulness in a respondent's life. The subscale consists of 5 items, and the total scores range between 5 and 35. Higher scores are indicative of better functioning and quality of life.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 22.51 (7.28) | 26.15 (8.78)

10. Secondary Outcome: Change in Perceived Level of Meaning in Life Using the Meaning in Life Questionnaire (MLQ)
Description: as for outcome 9
Time Frame: 6 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 33
score on a scale | 22.83 (9.03) | 25.55 (8.48)

11. Secondary Outcome: Change in Life Satisfaction Using the Satisfaction With Life Scale (SWLS)
Description: The SWLS is a measure of general satisfaction with one's life. Scores range from 5 to 35 with higher scores indicative of higher life satisfaction.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 20.83 (5.60) | 21.94 (6.90)

12. Secondary Outcome: Change in Life Satisfaction Using the Satisfaction With Life Scale (SWLS)
Description: as for outcome 11
Time Frame: 6 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 33
score on a scale | 20.83 (6.85) | 23.12 (7.69)

13. Secondary Outcome: Change in General Well-being Using the 5-item Version of the WHO Wellbeing Index (WBI-5)
Description: The WBI-5 measures participants' overall subjective well-being. Scores range between 0 and 15 with higher scores indicative of greater well-being.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 37
score on a scale | 8.26 (2.88) | 8.62 (2.58)

14. Secondary Outcome: Change in General Well-being Using the 5-item Version of the WHO Wellbeing Index (WBI-5)
Description: as for outcome 13
Time Frame: 6 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait-list Control Group
Number analyzed (Participants) | 35 | 33
score on a scale | 8.63 (2.70) | 9.27 (3.20)

15. Secondary Outcome: Perceived Negative Effects of the Intervention Using ad Hoc Questions
Description: Two questions were asked from respondents:
  1. "On the constellation seminar you participated in one month ago or since then, have you experienced any unfavorable change in your family life, your relationships with others or your interpersonal style in general that you attribute to the constellation seminar or can imagine that it is related to your participation in it?"
  2. "On the constellation seminar you participated in one month ago or since then, have you experienced any unfavorable mental or physical change in your personal life that you attribute to the constellation seminar or can imagine that it is related to your participation in it?" The number of participants who answered affirmatively to one or both questions above are reported here. Please note that the wording above is a hypersensitive approach to gather data on iatrogenic effects (cf. "can imagine that it is related to your participation").
Time Frame: 1 month post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 35
Participants | 13

16. Secondary Outcome: Perceived Negative Effects of the Intervention Using ad Hoc Questions
Description: Two questions were asked from respondents:
  1. "In the past 5 months (since the completion of the first follow-up questionnaire of this study), have you experienced any unfavorable change in your family life, your relationships with others or your interpersonal style in general that you attribute to the constellation seminar or can imagine that it is related to your participation in it?"
  2. "In the past 5 months (since the completion of the first follow-up questionnaire of this study), have you experienced any unfavorable mental or physical change in your personal life that you attribute to the constellation seminar or can imagine that it is related to your participation in it?" The number of participants who answered affirmatively to one or both questions above are reported here. Please note that the wording above is a hypersensitive approach to gather data on iatrogenic effects (cf. "can imagine that it is related to your participation").
Time Frame: 6 month post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 35
Participants | 9

ADVERSE EVENTS:
Time Frame: 1 month post-intervention
Description: Data on adverse events in the waitlist control group were unfortunately not collected due to a design flaw of this study.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 13/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=35)
Interpersonal relationships (Social circumstances) | 8 — Any unfavorable change in family life, relationships with others or interpersonal style in general
Any mild physical or mental health concern (General disorders) | 7 — Unfavorable mental or physical health change

LIMITATIONS AND CAVEATS:
* COVID-related changes in the intervention: 1) large reduction is dosage (8- instead of 16-24-hour workshop); 2) reduced group size (10 instead of the typical 20-25); 3) obligatory mask wearing influencing affect experiencing, expression, and recognition; 4) physical distancing requirements and subjective disease transmission risk perception decreasing engagement (intervention requires certain physical closeness).
* No adverse event data collected for control group.
* Low sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT05051462/Prot_SAP_ICF_000.pdf